CLINICAL TRIAL: NCT01487057
Title: "Evaluation of Lipid Metabolic Status and of Cardiovascular Risk at Patients With Thyroid Carcinoma, Radically Treated and With Chronic Thyroid Hormonal Substitution"
Brief Title: Lipid Metabolic Status in Thyroid Carcinoma
Acronym: LITCA
Status: Completed | Type: Observational
Sponsor: Prof. Dr. I. Chiricuta Institute of Oncology (Other)
Collaborators: Iuliu Hatieganu University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, PICIU DOINA, MD, PhD, Prof. Dr. I. Chiricuta Institute of Oncology
Other Study IDs: ChiricutaIO
Record Dates: First submitted 2011-12-05; First posted 2011-12-07 (Estimated); Last update posted 2012-12-27 (Estimated); Status verified 2012-12

CONDITIONS: Thyroid Carcinoma; Dyslipidemias; Risk Reduction Behavior; Hormone Replacement
Keywords: thyroid cancer; dislipidemia; cardiovascular risk
MeSH Terms: conditions — Thyroid Neoplasms; Dyslipidemias; Risk Reduction Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Thyroid cancer, lipids, LT4 withdrawal
- Thyroid cancer, Lipids, LT4 substitution

SUMMARY:
The continuous increase of the incidence of the thyroid cancer in the last years has taken this neoplasia among the first 4 frequent cancers in the cancer registry of the Institute of Oncology "Prof.Ion Chiricuţă" from Cluj-Napoca (IOCN), with a total number of over 470 new cases per year, added to the other 3700 cases already being in the evidence of the Institute.

The radical treatment brings for a long term a compensated chronic drug induces mYxoedema with it's important side effects. Among these one can find the dislipidemia and the change of the high sensitive C reactive protein (hsCRP) serological value. In the last years, many epidemiological studies have confirmed the fact that the patients with a high serological value of the hsCRP present a higher risk for the coronary disease and heart attack.

Prospective studies developed in european countries and in USA have provided results that are related to the predictive value of the hsCRP determinations over the cardiovascular risk. Thus, hsCRP is an indirect risk factor for the coronary disease. The risk for cardiovascular disease is 2 to 7 times higher at the people with a high level of hsCRP comparing to ones with low levels; the increase of the hsCRP serological value can be determined several years before the clinical debut of the coronary disease.

The screening for this population group with a high risk can introduce in use the prevention of the cardiac pathology and change the approach to the monitoring of the patients with thyroid cancer. A selection protocol will be elaborated for the patients that will withdraw the hormone treatment by using recombinant thyroid stimulating hormone (TSH) or will have personalised monitoring algorithm, with a shortening of the hormone treatment withdrawal.

DETAILED DESCRIPTION:
Although considered a rare type of cancer with an incidence under 6 cases for 100 000 persons, the thyroid carcinoma is the most frequent endocrine tumor. The incidence of this malignant disease has exponentially increased in the last decade, so that many specially centers in the world have focused on a better strategy of diagnosis, of treatment and of monitoring. By applying a suitable multimodal treatment, the prognosis of this disease is excellent, offering the patients a survival rate of over 90% at 10 years. During the monitoring of the disease, the patients are periodically supposed to withdraw the hormone treatment; because of this hormone imbalance, there will be important changes of the metabolism, especially the lipid one. This is the reason why we are preoccupied to increase the quality of life of the patients addicted to a chronic thyroid hormone therapy. The aim of this study is to demonstrate the way in which the lipid profile is influenced and to quantify the cardiovascular risk for the patients radically treated of thyroid cancer, by total thyroidectomy, metabolic irradiation and undergoing a chronic thyroid hormone treatment. Nowadays, Romania is one of the countries in which these patients are supposed to be kept in a iatrogenous myxoedema, the alternative being the recombinant thyroid stimulating hormone. For the patients with the mentioned diagnosis, the lipid profile will be determined and will consist of the following: total serologic cholesterol, cholesterol fractions, triglycerides and C reactive protein highly sensitive (hsCRP). A score for the cardiovascular accident risk will be elaborated. The attempt of classifying in cardiovascular risk groups the patients through the present study, would facilitate the selection of the patients and their access to therapies and modern monitoring strategies.

ELIGIBILITY:
Inclusion Criteria:

* thyroid carcinoma radically treated (surgery, radioiodine, thyroid hormone suppression )

Exclusion Criteria:

* other causes of high CRP (infection, inflammation)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will prospectively study a group of patients from the evidence of IOCN, with the histology of differentiated thyroid cancer, radically treated with total thyroidectomy, radioiodine therapy and undergoing chronic substitutive hormone treatment, levothyroxine. The evaluation of these patients will be done during the routine oncological control, after 6-12 months post therapy, while withdrawing the hormone treatment and inducing a short-term iatrogenic myxedema. We are estimating a total number of 30 patients with 3 successive determinations in 1 year. The ethics committee will evaluate this study and each patient will be included voluntarily, following clear information of the patient and an informed consent.
Sampling Method: Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2011-02; Primary Completion 2012-02 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
hsCRP an inflammatory biomarker for cardiovascular risk | May 2012
  hsCRP in thyroid hormone withdrwal for patients with thyroid carcinoma radically treated

SECONDARY OUTCOMES:
hsCRP may increase in repeated thyroid hormone withdrawal | May 2012

OTHER OUTCOMES:
hsCRP related to thyroid hormone withdrawal in patients with thyroid carcinoma radically treated | May 2012

CONTACTS AND LOCATIONS:
Overall Officials: Alexandru Irimie, PhD, Study Director — IOCN
Locations (1):
- Institute of Oncology "Prof.dr.I.Chiricuta", Cluj-Napoca, Cluj, Romania

REFERENCES:
- See also: Institute of Oncology "Prof.dr.i.Chiricuta" — http://www.iocn.ro
- See also: University of Medicine and Pharmacy "Iuliu Hatieganu" Cluj-Napoca — http://www.umfcluj.ro